CLINICAL TRIAL: NCT05063331
Title: Patient-Centered Outcomes of Sacrocolpopexy Versus Uterosacral Ligament Suspension for the Treatment of Uterovaginal Prolapse
Brief Title: Patient-Centered Outcomes in the Surgical Treatment of Uterovaginal Prolapse
Acronym: PREMIER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Case Western Reserve University (Other); MetroHealth Medical Center (Other); The Cleveland Clinic (Other); Duke University (Other); University of Pittsburgh (Other); Mayo Clinic (Other); Northwestern Medicine (Other)
Responsible Party: Principal Investigator, Adonis Hijaz, MD, Professor of Urology, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20210871
Record Dates: First submitted 2021-08-04; First posted 2021-10-01 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Uterine Prolapse
Keywords: Sacrocolpopexy; Uterosacral Ligament Suspension
MeSH Terms: conditions — Uterine Prolapse | interventions — Hysterectomy, Vaginal

STUDY DESIGN:
Intervention Model Description: The study is utilizing a 1:1 randomization scheme (by site) to assign patients to one of two treatment arms: 1) minimally invasive supracervical hysterectomy with sacrocolpopexy (MI-SCH+SCP, N=160) or 2) total vaginal hysterectomy with uterosacral ligament suspension (TVH+USLS, N=160).
Who Masked: Participant
Masking Description: Participants will be masked to the surgical randomization prior to surgery and will be informed of their surgical assignment (unmasked) after waking up from surgery and prior to discharge.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacrocolpopexy (Active Comparator): Minimally invasive supracervical hysterectomy with sacrocolpopexy (MI-SCH+SCP)
  Interventions: Procedure: Minimally invasive supracervical hysterectomy and sacrocolpopexy (MI-SCH+SCP)
- Uterosacral Ligament Suspension (Active Comparator): Total vaginal hysterectomy with uterosacral ligament suspension (TVH+USLS)
  Interventions: Procedure: Vaginal hysterectomy with uterosacral ligament suspension (TVH+USLS)

INTERVENTIONS:
Procedure: Minimally invasive supracervical hysterectomy and sacrocolpopexy (MI-SCH+SCP) — Minimally invasive robotic or laparoscopic supracervical hysterectomy will be done, and the vaginal apex (including cervix) will be suspended utilizing sacrocolpopexy mesh to the anterior spinous ligament.
  Arms: Sacrocolpopexy
Procedure: Vaginal hysterectomy with uterosacral ligament suspension (TVH+USLS) — The uterus will be removed vaginally and the vaginal apex will be suspended utilizing sutures in the uterosacral ligament.
  Arms: Uterosacral Ligament Suspension

SUMMARY:
The purpose of this study is to compare two types of surgery for the treatment of uterovaginal prolapse to determine which surgery works best from a patient's perspective and has the lowest number of short-term and long-term complications.

DETAILED DESCRIPTION:
This is a multi-site, randomized controlled trial, where women with the confirmed diagnosis of uterovaginal prolapse will be randomized in a 1:1 ratio to either A) a minimally invasive supracervical hysterectomy with sacrocolpopexy (MI-SCH+SCP) or B) total vaginal hysterectomy with uterosacral ligament suspension (TVH+USLS). After surgery, participants will be followed for 3 years including physical pelvic exams and validated symptom questionnaires to assess for the primary and secondary outcomes. A subset of participants will participate in semi-structured interviews, before surgery and through 2 years after surgery, that will assess patient recovery, satisfaction with care, and calibrate surveyed and clinically assessed outcomes to the daily life experiences of women.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥ 18 years of age and ≤ 80 years of age
2. Have diagnosis of symptomatic uterovaginal prolapse
3. Have elected to undergo surgical management of uterovaginal prolapse after consultation with their physician
4. Are eligible for both minimally invasive supracervical hysterectomy with sacrocolpopexy (MI-SCH+SCP) and total vaginal hysterectomy with uterosacral ligament suspension (TVH+USLS)

Exclusion Criteria:

1. Patients who wish to undergo uterine sparing procedures
2. Body mass index BMI) > 50
3. Previous hysterectomy or prior uterovaginal surgery
4. Have a diagnosis of neurogenic bladder, Parkinson's disease, multiple sclerosis, spinal cord injury, or cerebrovascular accident
5. Chronic indwelling urinary catheter
6. Urinary diversion of any type
7. Any condition or disorder that, in the opinion of the investigator, might prevent the subject from completing the study or interfere with the interpretation of the study results
8. Unable to speak, read, understand English

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | 36 months post-surgery
  The primary outcome is treatment failure defined as the presence of at least one of the following: 1) presence of a vaginal bulge defined as lead point of prolapse beyond the hymen, 2) report of bothersome vaginal bulge symptoms irrespective of stage of prolapse, or 3) retreatment of symptomatic prolapse with pessary, or surgery.

SECONDARY OUTCOMES:
Postoperative pain medication use | Post-surgery through Day 14
  Postoperative pain medication use will be assessed using the total morphine equivalent dosing (MED) for narcotics and using the total dosage for non-narcotics.
Change in surgical pain using VAS | Baseline, Days 1, 7 and 14 post-surgery
  Longitudinal pain score will be assessed using a visual analog scale (VAS) with a score of 0 to 100 where a higher score means a worse outcome.
Postoperative anti-emetic use | Post-surgery through Day 14
  Postoperative anti-emetic use will be assessed using the total number of times patients take an anti-emetic.
Change in nausea using VAS | Baseline, Days 1, 7 and 14 post-surgery
  Longitudinal nausea score will be assessed using a visual analog scale (VAS) with a score of 0 to 100 where a higher score means a worse outcome.
Change in fatigue using MAF | Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, and 8 post-surgery
  Fatigue will be assessed utilizing the Multi-Dimensional Assessment of Fatigue (MAF) Scale with a score of 1 to 148 where a higher score means a worse outcome.
Change in bladder function using UDI-6 | Baseline, 2, 6, 12, 24, and 36 months post-surgery
  Bladder function will be assessed using the Urinary Distress Inventory-6 (UDI-6) which is questions 15-20 of the Pelvic Floor Distress Inventory (PFDI-20) with a score of 0 to 18 where a higher score means a worse outcome.
Change in bladder function using IIQ-7 | Baseline, 2, 6, 12, 24, and 36 months post-surgery
  Bladder function will be assessed using the Incontinence Impact Questionnaire-7 (IIQ-7) with a score of 0 to 21 where a higher score means a worse outcome.
Change in bowel function using CRAD-8 | Baseline, 2, 6, 12, 24, and 36 months post-surgery
  Bowel function will be assessed using the Colorectal Anal Distress Inventory 8 (CRAD-8) which is questions 7-14 of the Pelvic Floor Distress Inventory (PFDI-20) with a score of 0 to 24 where a higher score means a worse outcome.
Change in sexual function using PISQ-12 | Baseline, 6, 12, 24, and 36 months post-surgery
  Sexual function will be assessed using the Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) with a score of 0 to 48 where a higher score means a worse outcome.
Change in sexual function using FSFI | Baseline, 6, 12, 24, and 36 months post-surgery
  Sexual function will be assessed using the Female Sexual Function Inventory (FSFI) with a score of 2 to 36 where higher score where a higher score means a better outcome.
Change in body image using BIPOP | Baseline, 6, 12, 24, and 36 months post-surgery
  Body image will be assessed using the Body Image in Pelvic Organ Prolapse Questionnaire (BIPOP) with a score of 1 to 5 where a higher score means a better outcome.
Change in quality of life using P-QOL | Baseline, 2, 6, 12, 24, and 36 months post-surgery
  General quality of life will be assessed using the Pelvic Organ Prolapse Quality of Life Questionnaire (P-QOL) with a score in each domain of 0 to 100 where a higher score means a worse outcome.
Change in satisfaction with care using PGI-I | Baseline, 6, 12, 24, and 36 months post-surgery
  Satisfaction with care will be assessed using the Patient Global Impression of Improvement (PGI-I) scale with a score of 1 to 7 where higher score means a worse outcome.
Rate of Grade I-V DINDO complications in each surgical arm | Surgery through 36 months post-surgery
  Surgical complications will be assessed using the Clavien-Dindo standardized classification system with a grade of I to V where the higher grade means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Adonis Hijaz, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (7):
- United States (7):
  - Mayo Clinic, Jacksonville, Florida
  - Northwestern Medicine, Chicago, Illinois
  - Duke University, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh, UPMC Magee-Womens Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be made available after de-identification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 9 months and ending 36 months following publication.
Access Criteria: Researchers who provide a methodologically sound proposal may use the data for any purpose.